CLINICAL TRIAL: NCT00998296
Title: Phase I Dose Escalation Study of Concomitant BIBF 1120 and BIBW 2992 in Patients With Advanced Solid Tumours.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1239.14; 2009-011321-14 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib; nintedanib

ARMS (1):
- BIBW 2992 + BIBF 1120 (Experimental): This is a phase I dose escalation clinical trial and the data obtained shall determine the MTD for the combination of BIBW 2992/BIBF 1120 in 28-day of treatment.
  Interventions: Drug: BIBW 2992; Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBW 2992 — EGFR inhibitor
Drug: BIBF 1120 — VEGF inhibitor

SUMMARY:
The primary objective of this trial is to determine the Maximum Tolerated Dose (MTD) of the combination of BIBW 2992/BIBF 1120 therapy administered concomitantly. The MTD will provide dosing recommendation for subsequent phase II trials in patients with metastatic cancer.

ELIGIBILITY:
Inclusion criteria:

1. Patients with confirmed histological or cytological diagnosis of advanced solid tumours and for whom no proven therapy exists or who are not amenable to established treatments.
2. Age 18 years or older.
3. Life expectancy of at least three months.
4. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
5. Patients previously treated and with asymptomatic brain metastases are eligible
6. Patients must have recovered from recent surgery.

Exclusion criteria:

1. Active infectious disease
2. Recent surgery within the last 4 weeks prior visit 1.
3. Chronic diarrhoea or gastrointestinal tract disease resulting in an inability to take oral medication
4. History of haemorrhagic or thrombotic events
5. Significant cardiovascular diseases within
6. Current peripheral neuropathy > Common Terminology Criteria for Adverse Events (CTCAE) grade 1 except due to trauma
7. Untreated or symptomatic brain metastases or leptomeningeal disease.
8. Treatment with an Epidermal growth Factor-receptor (EGFR)- or Heregulin Receptor 2 (HER2) inhibiting drug or antiangiogenic drug.
9. Therapeutic anticoagulation.
10. Female patients of childbearing potential.
11. Known pre-existing interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1239.14.3301A Boehringer Ingelheim Investigational Site, Villejuif, France

REFERENCES:
- [Derived] Bahleda R, Hollebecque A, Varga A, Gazzah A, Massard C, Deutsch E, Amellal N, Farace F, Ould-Kaci M, Roux F, Marzin K, Soria JC. Phase I study of afatinib combined with nintedanib in patients with advanced solid tumours. Br J Cancer. 2015 Nov 17;113(10):1413-20. doi: 10.1038/bjc.2015.374. Epub 2015 Oct 29. PMID 26512876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial consisted of a dose-escalation phase (to determine the maximum tolerated dose (MTD) of treatments administered concomitantly) and an expansion phase(to assess the safety and the preliminary anti-tumour activity of the combination therapy at the previously determined MTD in patients with non-small cell lung cancer or pancreatic adenocarcinoma)
Groups:
- Nintedanib 150 mg +Afatinib 30 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 150 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 30 mg was given continuously once daily (q.d.).
  This is a part of the "dose-escalation phase".
- Nintedanib 150 mg +Afatinib 40 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 150 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 40 mg was given continuously once daily (q.d.).
  This is a part of the "dose-escalation phase".
- Nintedanib 200 mg +Afatinib 10 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 10 mg was given continuously once daily (q.d.).
  This is a part of the "dose-escalation phase".
- Nintedanib 200 mg +Afatinib 20 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 20 mg was given continuously once daily (q.d.).
  This is a part of the "dose-escalation phase".
- Nintedanib 200 mg +Afatinib 30 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 30 mg was given continuously once daily (q.d.).
  This is a part of the "dose-escalation phase".
- Nintedanib 200 mg +Afatinib 40 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 40 mg was given continuously once daily (q.d.).
  This is a part of the "dose-escalation phase".
- Nintedanib 150 mg +Afatinib 40 mg - Intermittently: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 150 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 40 mg was given intermittently once daily (q.d.) every other week.
  This is a part of the "dose-escalation phase".
- Nintedanib 200 mg +Afatinib 30 mg - Intermittently: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 30 mg was given intermittently once daily (q.d.) every other week.
  This is a part of the "dose-escalation phase".
- Nintedanib 200 mg +Afatinib 40 mg - Intermittently: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 40 mg was given intermittently once daily (q.d.) every other week.
  This is a part of the "dose-escalation phase".
- NSCLC: Patients with non-small cell lung cancer (NSCLC) receiving the study drug combination at the maximum tolerated dose (MTD) level determined for continuous afatinib and nintedanib dosing during the dose-escalation phase (oral administration of soft-gelatine capsule of Nintedanib 150 mg (b.i.d.) plus film-coated tablet of Afatinib 30 mg (q.d.)).
  This is a part of the "expansion phase" which follows on the dose-escalation phase.
- Pancreatic Adenocarcinoma: Patients with Pancreatic adenocarcinoma were to be treated with the study drug combination at the maximum tolerated dose (MTD) level determined for continuous afatinib and nintedanib dosing during the dose-escalation phase (oral administration of soft-gelatine capsule of Nintedanib 150 mg bid plus film-coated tablet of Afatinib 30 mg qd).
  This is a part of the "expansion phase" which follows on the dose-escalation phase.
Period: Overall Study
Arm/Group | Nintedanib 150 mg +Afatinib 30 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Continuously | Nintedanib 200 mg +Afatinib 10 mg - Continuously | Nintedanib 200 mg +Afatinib 20 mg - Continuously | Nintedanib 200 mg +Afatinib 30 mg - Continuously | Nintedanib 200 mg +Afatinib 40 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Intermittently | Nintedanib 200 mg +Afatinib 30 mg - Intermittently | Nintedanib 200 mg +Afatinib 40 mg - Intermittently | NSCLC | Pancreatic Adenocarcinoma
Started | 6 | 3 | 3 | 3 | 8 | 3 | 7 | 6 | 6 | 18 | 7
Completed | 6 (Did not discontinue treatment before or at Day 28) | 2 (Did not discontinue treatment before or at Day 28) | 3 (Did not discontinue treatment before or at Day 28) | 3 (Did not discontinue treatment before or at Day 28) | 6 (Did not discontinue treatment before or at Day 28) | 3 (Did not discontinue treatment before or at Day 28) | 6 (Did not discontinue treatment before or at Day 28) | 4 (Did not discontinue treatment before or at Day 28) | 4 (Did not discontinue treatment before or at Day 28) | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 2 | 18 | 7
Not completed — Progressive disease | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 14 | 5
Not completed — Dose limiting or dose reducing toxicity | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Other adverse event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Refused to continue taking trial med. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Reason other than those specified above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): A treated set (TS) was defined consisting of all patients who received at least one dose of nintedanib or afatinib during the study period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib 150 mg +Afatinib 30 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Continuously | Nintedanib 200 mg +Afatinib 10 mg - Continuously | Nintedanib 200 mg +Afatinib 20 mg - Continuously | Nintedanib 200 mg +Afatinib 30 mg - Continuously | Nintedanib 200 mg +Afatinib 40 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Intermittently | Nintedanib 200 mg +Afatinib 30 mg - Intermittently | Nintedanib 200 mg +Afatinib 40 mg - Intermittently | NSCLC | Pancreatic Adenocarcinoma | Total
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 8 | 3 | 7 | 6 | 6 | 18 | 7 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (8.1) | 51.7 (1.5) | 46.7 (4.9) | 53.3 (11.0) | 51.5 (9.7) | 44.3 (8.1) | 64.9 (3.5) | 52.2 (6.0) | 63.3 (10.3) | 58.1 (10.9) | 58.1 (6.8) | 56.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 1 | 6 | 2 | 0 | 4 | 2 | 11 | 1 | 31
  Male | 3 | 2 | 3 | 2 | 2 | 1 | 7 | 2 | 4 | 7 | 6 | 39

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Nintedanib and Afatinib Based on the Percentage of Participants Experienced Dose Limiting Toxicities
Description: Maximum tolerated dose (MTD) of nintedanib and afatinib based on the Percentage of participants experienced dose limiting toxicities during the dose escalation phase.
Time Frame: first treatment cycle, up to 28 days
Population: TS
Measure: Number; unit: percentage of participants
Arm/Group | Nintedanib 150 mg +Afatinib 30 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Continuously | Nintedanib 200 mg +Afatinib 10 mg - Continuously | Nintedanib 200 mg +Afatinib 20 mg - Continuously | Nintedanib 200 mg +Afatinib 30 mg - Continuously | Nintedanib 200 mg +Afatinib 40 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Intermittently | Nintedanib 200 mg +Afatinib 30 mg - Intermittently | Nintedanib 200 mg +Afatinib 40 mg - Intermittently
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 8 | 3 | 7 | 6 | 6
percentage of participants
  Alanine aminotransferase increased | 0.0 | 0.0 | 0.0 | 0.0 | 12.5 | 33.3 | 0.0 | 0.0 | 0.0
  Aspartate aminotransferase increased | 0.0 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0 | 0.0 | 0.0 | 0.0
  Blood creatinine increased | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 0.0 | 16.7 | 0.0
  Dehydration | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7
  Diarrhoea | 0.0 | 33.3 | 0.0 | 0.0 | 25.0 | 33.3 | 0.0 | 16.7 | 0.0
  Hepatocellular injury | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 0.0 | 16.7 | 0.0
  Renal failure acute | 0.0 | 66.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Hepatotoxicity | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7

2. Secondary Outcome: Overall Tumour Response Rate Assessed by the Investigator According to the Response Evaluation Criteria In Solid Tumours (RECIST) Version 1.1
Description: The investigator evaluated whether complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD) occurred in a patient.
  CR for target lesions: Disappearance of all target lesions. CR for non-target lesions: Disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10mm short axis).
  PR: At least a 30% decrease in the sum of diameters (SoD) of target lesions taking as reference the baseline sum diameters.
  SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as references the smallest SoD while on study.
  PD: At least a 20% increase in the SoD of target lesions, taking as references the smallest sum on study (this includes the baseline sum if that is the smallest on study). Also, the sum must also demonstrate an absolute increase of a least 5mm. Appearance of one or more new lesions
Time Frame: 6 weeks
Population: TS
Measure: Number; unit: percentage of participants
Arm/Group | Nintedanib 150 mg +Afatinib 30 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Continuously | Nintedanib 200 mg +Afatinib 10 mg - Continuously | Nintedanib 200 mg +Afatinib 20 mg - Continuously | Nintedanib 200 mg +Afatinib 30 mg - Continuously | Nintedanib 200 mg +Afatinib 40 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Intermittently | Nintedanib 200 mg +Afatinib 30 mg - Intermittently | Nintedanib 200 mg +Afatinib 40 mg - Intermittently | NSCLC | Pancreatic Adenocarcinoma
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 7 | 3 | 6 | 6 | 3 | 17 | 6
percentage of participants
  Complete response | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Partial response | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 17.6 | 0.0
  Stable disease | 66.7 | 66.7 | 66.7 | 33.3 | 71.4 | 100 | 66.7 | 83.3 | 100.0 | 70.6 | 33.3
  Progressive disease | 33.3 | 33.3 | 33.3 | 66.7 | 28.6 | 0.0 | 33.3 | 16.7 | 0.0 | 11.8 | 66.6

3. Secondary Outcome: Incidence and Intensity of Adverse Events According to CTCAE (Common Toxicity Criteria Adverse Event) Version 3.0
Description: Incidence and intensity of Adverse Events with grading according to the Common Terminology Criteria for Adverse Events (CTCAE version 3.0).
Time Frame: First treatment administration until cut-off date of 02Oct2014; up to 336 days
Population: TS
Measure: Number; unit: participants
Arm/Group | Nintedanib 150 mg +Afatinib 30 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Continuously | Nintedanib 200 mg +Afatinib 10 mg - Continuously | Nintedanib 200 mg +Afatinib 20 mg - Continuously | Nintedanib 200 mg +Afatinib 30 mg - Continuously | Nintedanib 200 mg +Afatinib 40 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Intermittently | Nintedanib 200 mg +Afatinib 30 mg - Intermittently | Nintedanib 200 mg +Afatinib 40 mg - Intermittently | NSCLC | Pancreatic Adenocarcinoma
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 8 | 3 | 7 | 6 | 6 | 18 | 7
participants
  CTCAE Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  CTCAE Grade 2 | 2 | 0 | 1 | 2 | 1 | 0 | 2 | 4 | 0 | 7 | 2
  CTCAE Grade 3 | 1 | 2 | 2 | 1 | 5 | 2 | 4 | 2 | 3 | 7 | 2
  CTCAE Grade 4 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 2
  CTCAE Grade 5 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0

4. Secondary Outcome: Changes in Safety Laboratory Parameters
Description: Changes in safety laboratory Parameters reported as adverse events
Time Frame: First treatment administration until cut-off date of 02 October 2014, up to 336 days
Population: TS
Measure: Number; unit: participants
Arm/Group | Nintedanib 150 mg +Afatinib 30 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Continuously | Nintedanib 200 mg +Afatinib 10 mg - Continuously | Nintedanib 200 mg +Afatinib 20 mg - Continuously | Nintedanib 200 mg +Afatinib 30 mg - Continuously | Nintedanib 200 mg +Afatinib 40 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Intermittently | Nintedanib 200 mg +Afatinib 30 mg - Intermittently | Nintedanib 200 mg +Afatinib 40 mg - Intermittently | NSCLC | Pancreatic Adenocarcinoma
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 8 | 3 | 7 | 6 | 6 | 18 | 7
participants
  Alanine aminotransferase increased | 1 | 1 | 1 | 1 | 3 | 3 | 1 | 3 | 3 | 1 | 1
  Aspartate aminotransferase increased | 1 | 1 | 1 | 0 | 3 | 3 | 1 | 2 | 1 | 1 | 2
  Blood creatinine increased | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0
  Blood alkaline phosphatase increased | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Blood bilirubin increased | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Troponin increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
  Blood creatinine phosphokinase increased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood fibrinogen increased | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hepatic enzymes increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Cpre,ss,Norm (Dose Normalized Trough Plasma Concentration of Nintedanib at Steady State)
Description: Cpre,ss,norm (Dose normalized trough plasma concentration of nintedanib at steady state) are presented for the 2 MTD treatment groups (continuous administered nintedanib at 150 mg b.i.d. concomitantly with continuously administered afatinib 30 mg q.d. or with intermittently administered afatinib 40 mg q.d.)
  As nintedanib is given twice daily, samples are taken at Day 8, Day 15, Day 22 and Day 28; the Pharmacokinetic (PK) parameter names will be Cpre,ss,15,norm (Day 8), Cpre,ss,29,norm (Day 15), Cpre,ss,43,norm (Day 22) and Cpre,ss,55,norm (Day 28)
Time Frame: Day 8, Day 15, Day 22 and Day 28
Population: PKS. Only 6 patients were planned to be treated in the "Nintedanib 150 mg +Afatinib 30 mg- Continuously" group. Nevertheless, the patients were allowed to reduce their dose and by the way they changed the group and came in the "Nintedanib 150 mg +Afatinib 30 mg- Continuously" group with at the end N = 8 evaluable concentrations instead of 6 planned
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/millilitre/milligram (ng/mL/mg)
Groups:
- Nintedanib 150 mg +Afatinib 30 mg- Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 150 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 30 mg was given continuously once daily (q.d.).
  This is a part of the "dose-escalation phase".
- Nintedanib 150 mg +Afatinib 40 mg- Intermittently: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 150 mg continuously twice daily (b.i.d.); concomitantly, film-coated tablet of Afatinib 40 mg was given intermittently once daily (q.d.) every other week.
  This is a part of the "dose-escalation phase".
Arm/Group | Nintedanib 150 mg +Afatinib 30 mg- Continuously | Nintedanib 150 mg +Afatinib 40 mg- Intermittently
Number analyzed (Participants) | 8 | 7
nanogram/millilitre/milligram (ng/mL/mg)
  Cpre,ss,15,norm (N= 6, 7) | 0.122 (155) | 0.0731 (92.2)
  Cpre,ss,29,norm (N= 6, 6) | 0.0948 (136) | 0.0755 (148)
  Cpre,ss,43,norm (N= 5, 6) | 0.112 (125) | 0.0762 (79.7)
  Cpre,ss,55,norm (N= 8, NA) | 0.0797 (247) | NA (NA) — Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

6. Secondary Outcome: Trough Plasma Concentration of Afatinib at Steady State
Description: C(pre,ss) is defined as pre-dose (trough) concentration of afatinib in plasma at steady state immediately before administration of the next dose.
  C24,7 corresponds to the plasma concentration at 24 hours on Day 7. C24,13 corresponds to the plasma concentration at 24 hours on Day 13. C24,27 corresponds to the plasma concentration at 24 hours on Day 27.
Time Frame: Day 7, Day 13, Day 15, Day 22, Day 27 and Day 28
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/millilitre (ng/mL)
Arm/Group | Nintedanib 150 mg +Afatinib 30 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Intermittently
Number analyzed (Participants) | 8 | 7
nanogram/millilitre (ng/mL)
  Cpre,ss,15 (N= 6, NA) | 15.5 (62.0) | NA (NA) — Not applicable (Value not calculated): Cpre,ss,15 was calculated for the intermittent treatment because the values were not available. No blood was taken at this time
  Cpre,ss,22 (N= 6, NA) | 19.0 (56.5) | NA (NA) — Not applicable (Value not calculated): Cpre,ss,22 was calculated for the intermittent treatment because the values were not available. No blood was taken at this time
  Cpre,ss,28 (N= 8, NA) | 19.1 (63.3) | NA (NA) — Not applicable (Value not calculated): Cpre,ss,28 was calculated for the intermittent treatment because the values were not available. No blood was taken at this time
  C24,7 (N= NA, 6) | NA (NA) — Not applicable (Value not calculated): C24,7 was calculated for the intermittent treatment; So, not available for the first treatment because no blood was taken at this time | 19.6 (127.0)
  C24,13 (N= NA, 5) | NA (NA) — Not applicable (Value not calculated): C24,13 was calculated for the intermittent treatment; So, not available for the first treatment because no blood was taken at this time | 11.5 (76.4)
  C24,27 (N= NA, 2) | NA (NA) — Not applicable (Value not calculated): C24,27 was calculated for the intermittent treatment; So, not available for the first treatment because no blood was taken at this time | 30.5 (21.9)

7. Secondary Outcome: Objective Response (OR) During the Expansion Phase
Description: OR is defined as a best overall response of complete response (CR) or partial response (PR) according to RECIST version 1.1, CR for target lesions (TL): Disappearance of all target lesions.
  CR for non-target lesions (NTL): Disappearance of all non-target lesions. All lymph nodes must be nonpathological in size (<10mm short axis). PR for TL: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
  Other factors which add to the overall response of an imaging timepoint as PR are as below:
  CR in TL, but non-CR/Non-PD in NTL leads to PR CR in TL, but not evaluated NTL leads to PR PR in TL, but non-PD NTL or not all evaluated NTL leads to PR; All the above scenarios should also satisfy 'No occurrence of new lesions'.
Time Frame: Tumour assessment was to be performed at Screening, every 6 weeks after starting study treatment until disease progression, and at the end-of-treatment (EOT) visit (up to 1117 days)
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC | Pancreatic Adenocarcinoma
Number analyzed (Participants) | 18 | 7
percentage of participants
  Yes | 22.2 | 0.0
  No | 72.2 | 85.7
  Missing | 5.6 | 14.3

8. Secondary Outcome: Disease Control (DC) During the Expansion Phase
Description: DC is defined as the best overall response of CR, PR, stable disease (SD) and non-CR/non-PD. CR for target lesions (TL): Disappearance of all target lesions. CR for non-target lesions (NTL): Disappearance of all non-target lesions . All lymph nodes must be non-pathological in size (<10mm short axis). PR for TL: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. Other factors which add to the overall response of an imaging timepoint as PR are as below:- CR in TL, but non-CR/Non-PD in NTL leads to PR CR in TL, but not evaluated NTL leads to PR PR in TL, but non-PD NTL or not all evaluated NTL leads to PR; SD for TL: change in the sum of diameters does not satisfy PR or PD. SD in TL, non-PD in NTL lead to overall response of SD, provided there is no appearance of new lesions.
Time Frame: as for outcome 7
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC | Pancreatic Adenocarcinoma
Number analyzed (Participants) | 18 | 7
percentage of participants
  Yes | 83.3 | 28.6
  No | 11.1 | 57.1
  Missing | 5.6 | 14.3

9. Secondary Outcome: Stable Disease for at Least 12 Weeks During the Expansion Phase
Description: SD: Neither sufficient shrinkage to qualify for PR (Partial response) nor sufficient increase to qualify for PD(Progressive disease), taking as references the smallest sum of diameters SoD while on study.
  PR: At least a 30% decrease in the sum of diameters (SoD) of target lesions taking as reference the baseline sum diameters.
  PD: At least a 20% increase in the SoD of target lesions, taking as references the smallest sum on study (this includes the baseline sum if that is the smallest on study). Also, the sum must also demonstrate an absolute increase of a least 5mm. Appearance of one or more new lesions.
Time Frame: as for outcome 7
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC | Pancreatic Adenocarcinoma
Number analyzed (Participants) | 18 | 7
percentage of participants
  Yes | 44.4 | 0.0
  No | 50.0 | 85.7
  Missing | 5.6 | 14.3

10. Secondary Outcome: Percentage Change in the Tumour Size From Baseline During the Expansion Phase
Description: Percentage change in the tumour size from baseline is expressed as Number of subjects with maximum decrease from baseline in the sum of longest diameters of target lesions.
Time Frame: as for outcome 7
Population: Treated set
Measure: Number; unit: participants
Arm/Group | NSCLC | Pancreatic Adenocarcinoma
Number analyzed (Participants) | 16 | 6
participants
  >=20% | 1 | 3
  >=0% and <20% | 4 | 3
  >-30% and <0% | 6 | 0
  <-30% | 5 | 0

ADVERSE EVENTS:
Time Frame: First treatment administration until cut-off date of 02Oct2014; up to 336 days
Groups:
- Nintedanib 150 mg +Afatinib 30 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 150 mg continuously twice daily (b.i.d.); concomitantly, filmcoated tablet of Afatinib 30 mg was given continuously once daily (q.d.)
- Nintedanib 150 mg +Afatinib 40 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 150 mg continuously twice daily (b.i.d.); concomitantly, filmcoated tablet of Afatinib 40 mg was given continuously once daily (q.d.)
- Nintedanib 200 mg +Afatinib 10 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, filmcoated tablet of Afatinib 10 mg was given continuously once daily (q.d.)
- Nintedanib 200 mg +Afatinib 20 mg - Continuosly: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, filmcoated tablet of Afatinib 20 mg was given continuously once daily (q.d.)
- Nintedanib 200 mg +Afatinib 30 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, filmcoated tablet of Afatinib 30 mg was given continuously once daily (q.d.)
- Nintedanib 200 mg +Afatinib 40 mg - Continuously: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, filmcoated tablet of Afatinib 40 mg was given continuously once daily (q.d.)
- Nintedanib 150 mg +Afatinib 40 mg - Intermittently: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 150 mg continuously twice daily (b.i.d.); concomitantly, filmcoated tablet of Afatinib 40 mg was given intermittently once daily (q.d.) every other week
- Nintedanib 200 mg +Afatinib 30 mg - Intermittently: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, filmcoated tablet of Afatinib 30 mg was given intermittently once daily (q.d.) every other week
- Nintedanib 200 mg +Afatinib 40 mg - Intermittently: Patients receiving oral administration of soft-gelatine capsule of Nintedanib 200 mg continuously twice daily (b.i.d.); concomitantly, filmcoated tablet of Afatinib 40 mg was given intermittently once daily (q.d.) every other week
- Pancreatic Adenocarcinoma: Patients with Pancreatic adenocarcinoma were to be treated with the study drug combination at the maximum tolerated dose (MTD) level determined for continuous afatinib and nintedanib dosing during the dose-escalation phase (oral administration of soft-gelatine capsule of Nintedanib 150 mg (b.i.d) plus film-coated tablet of Afatinib 30 mg (q.d)). This is a part of the "expansion phase" which follows on the dose-escalation phase.
Arm/Group | Nintedanib 150 mg +Afatinib 30 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Continuously | Nintedanib 200 mg +Afatinib 10 mg - Continuously | Nintedanib 200 mg +Afatinib 20 mg - Continuosly | Nintedanib 200 mg +Afatinib 30 mg - Continuously | Nintedanib 200 mg +Afatinib 40 mg - Continuously | Nintedanib 150 mg +Afatinib 40 mg - Intermittently | Nintedanib 200 mg +Afatinib 30 mg - Intermittently | Nintedanib 200 mg +Afatinib 40 mg - Intermittently | NSCLC | Pancreatic Adenocarcinoma
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/3 | 1/3 | 0/3 | 7/8 | 3/3 | 1/7 | 1/6 | 4/6 | 7/18 | 3/7
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 3/3 | 8/8 | 3/3 | 7/7 | 6/6 | 6/6 | 18/18 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 150 mg +Afatinib 30 mg - Continuously (N=6) | Nintedanib 150 mg +Afatinib 40 mg - Continuously (N=3) | Nintedanib 200 mg +Afatinib 10 mg - Continuously (N=3) | Nintedanib 200 mg +Afatinib 20 mg - Continuosly (N=3) | Nintedanib 200 mg +Afatinib 30 mg - Continuously (N=8) | Nintedanib 200 mg +Afatinib 40 mg - Continuously (N=3) | Nintedanib 150 mg +Afatinib 40 mg - Intermittently (N=7) | Nintedanib 200 mg +Afatinib 30 mg - Intermittently (N=6) | Nintedanib 200 mg +Afatinib 40 mg - Intermittently (N=6) | NSCLC (N=18) | Pancreatic Adenocarcinoma (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 150 mg +Afatinib 30 mg - Continuously (N=6) | Nintedanib 150 mg +Afatinib 40 mg - Continuously (N=3) | Nintedanib 200 mg +Afatinib 10 mg - Continuously (N=3) | Nintedanib 200 mg +Afatinib 20 mg - Continuosly (N=3) | Nintedanib 200 mg +Afatinib 30 mg - Continuously (N=8) | Nintedanib 200 mg +Afatinib 40 mg - Continuously (N=3) | Nintedanib 150 mg +Afatinib 40 mg - Intermittently (N=7) | Nintedanib 200 mg +Afatinib 30 mg - Intermittently (N=6) | Nintedanib 200 mg +Afatinib 40 mg - Intermittently (N=6) | NSCLC (N=18) | Pancreatic Adenocarcinoma (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 4 | 0 | 0 | 2 | 1 | 4 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Aerophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 3 | 3 | 8 | 3 | 6 | 6 | 6 | 14 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 2 | 3 | 4 | 2 | 4 | 3 | 5 | 12 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tongue dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 5 | 3 | 3 | 5 | 5 | 6 | 0
Asthenia (General disorders) | 6 | 3 | 2 | 3 | 8 | 3 | 5 | 2 | 3 | 13 | 2
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal dryness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 2 | 0 | 1 | 0 | 2 | 0 | 1 | 3 | 5 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Oedema peripheral (General disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 2 | 1 | 2 | 0 | 0 | 2 | 2 | 1 | 1
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 4 | 2 | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iodine allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 4 | 3 | 0 | 2 | 4 | 1 | 4 | 2 | 3 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Purulent discharge (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 1 | 3 | 3 | 4 | 2 | 1 | 0 | 2 | 5 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 3 | 3 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 2 | 3 | 1 | 2 | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 1 | 2 | 3 | 3 | 4 | 6 | 4 | 11 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 2 | 3 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 2 | 2 | 1 | 2 | 1 | 2 | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 5 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical root pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0
Parosmia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0
Expressive language disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Libido disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Psychomotor retardation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 3 | 0 | 1 | 1 | 2 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 3 | 0 | 1 | 2 | 2 | 1 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 3 | 5 | 2 | 1 | 0 | 2 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2 | 4 | 1 | 3 | 3 | 0 | 5 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 11 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 5 | 1 | 0 | 0 | 0 | 5 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Statistics of PK parameters are only estimated when at least 2/3 of the data are evaluable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.